CLINICAL TRIAL: NCT00613028
Title: Phase II Study of Bevacizumab Plus Either Temozolomide or Etoposide for (GBM) Patients Who Have Failed Bevacizumab Plus Irinotecan
Brief Title: Ph II Bev + Either Temozolomide/Etoposide for GBM Pts Who Have Failed Bev + Irinotecan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003768
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; GBM; Bevacizumab; Avastin; Etoposide; Brain tumor; Irinotecan; Glioblastoma multiforme; Temodar; Temozolomide; Etopophos; Toposar; VePesid; VP-16; Camptosar
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bevacizumab; Temozolomide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temo + Avastin (Experimental): Patients treated with bevacizumab + temozolomide
  Interventions: Drug: Temo + Avastin
- VP-16 + Avastin (Experimental): Patients treated with bevacizumab and VP-16 (etoposide)
  Interventions: Drug: VP-16 + Avastin

INTERVENTIONS:
Drug: Temo + Avastin — Patients have progressed/had gr3/> toxicity related to etoposide, with no had progression/gr 3/> toxicity related to temozolomide, will only be considered for bevacizumab and temozolomide. Bevacizumab intravenously at dose 10mg/kg every other wk. For patients on bevacizumab and temozolomide, temozolomide administered on continuous dosing schedule at 50mg/m2/day.
  Other Names: temozolomide; temodar; bevacizumab
  Arms: Temo + Avastin
Drug: VP-16 + Avastin — Patients have progressed/had gr3/> toxicity related to temozolomide, but have not progressed/gr3/> toxicity related to etoposide,considered only for bevacizumab and etoposide. Bevacizumab intravenously at dose 10mg/kg every other wk. Patients on bevacizumab and etoposide, etoposide once daily at 50mg/m2/day first 21 days of each 28-day cycle.
  Other Names: VP-16; etoposide; bevacizumab; avastin
  Arms: VP-16 + Avastin

SUMMARY:
Primary objective To estimate 6-month progression free survival probability of pts w recurrent GBM treated w bev + either daily temozolomide/etoposide following progression on bev + irinotecan Secondary Objectives To evaluate safety & tolerability of bev + either daily temozolomide/etoposide among pts w recurrent GBM who have progressed on bev + irinotecan To evaluate radiographic response, progression free survival & overall survival of pts w recurrent GBM treated w bev + either daily temozolomide/etoposide following progression on bev + irinotecan

DETAILED DESCRIPTION:
This is exploratory, two-arm, phase II study designed to assess anti-tumor activity of bev + either daily temozolomide/etoposide among GBM pts w progressive disease following bev + irinotecan. About 48 participants w recurrent GBM will take part in this study. Approximately 24 participants will receive bev plus temozolomide & approximately 24 will receive bev + etoposide. Pts must have confirmed diagnosis of GBM & radiographic evidence of recurrence following prior therapy bev + irinotecan. 24 pts will be enrolled onto each arm of this single-stage study. If 4 or more of these 24 pts live 6/more months without disease progression, treatment regimen will be considered worthy of further investigation. Otherwise, treatment regimen will be determined not worthy of further investigation within pt population. Type I & II error rates associated w testing are 0.030 & 0.115 respectively. Management guidelines dose reduction/interruption for temo, etoposide, & bev.

ELIGIBILITY:
Inclusion Criteria:

* Pts have confirmed diagnosis of GBM & radiographic evidence of recurrence following prior therapy w bev + irinotecan
* Age >18 yrs
* Interval of >4 wks between prior surgical resection/1 week from stereotactic biopsy
* Interval of >12 wks from end of prior external beam radiation therapy (XRT) unless there is new area of enhancement consistent w recurrent tumor outside of XRT field,/there are progressive changes on MRI on >2 consecutive MRI scans >4wks apart, /there is biopsy-proven tumor progression
* Interval of >4 wks from prior chemo / investigational agent unless pt has recovered from all anticipated toxicities associated w that therapy.
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Hematocrit >29percent, absolute neutrophil count (ANC)>1,000 cells/ml l, platelets > 100,000 cells/ml l
* Serum creatinine<1.5 mg/dl, serum glutamate oxaloacetate transaminase (SGOT) & bilirubin<1.5 times upper limit of normal (ULN)
* Signed informed consent approved by Institutional Review Board (IRB) prior to pt entry
* No evidence of hemorrhage on baseline MRI/CT scan other than those that are stable gr1
* If sexually active, pts will take contraceptive measures for duration of treatments

Exclusion Criteria:

* Co-medication that may interfere w study results
* Active infection requiring intravenous antibiotics
* Progression to daily etoposide/progression to daily temo
* Gr3/greater toxicity related to prior bev therapy,/prior temozolomide/etoposide
* Requires therapeutic anti-coagulation with warfarin.
* Inability to comply w study and/or follow-up procedures
* Current, recent,/planned participation in experimental drug study other than Genentech-sponsored bev cancer study
* Inadequately controlled hypertension
* Any prior history of hypertensive crisis/hypertensive encephalopathy
* New York Heart Association (NYHA) Gr II/greater congestive heart failure
* History of myocardial infarction (MI)/unstable angina within 6 mths prior to study enrollment
* History of stroke/transient ischemic attack within 6 mths prior to study enrollment
* Significant vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either:
* urine protein:creatinine (UPC) ratio >1.0 at screening /
* Urine dipstick for proteinuria ≥ 2+
* Known hypersensitivity to any component of bevacizumab
* Pregnant or lactating. Use of effective means of contraception in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide Arm: Bevacizumab + Temozolomide: Patients who progressed or had grade 3 or greater toxicity related to prior daily etoposide dosing, but have not had prior progression or grade 3 toxicity related to prior daily temozolomide therapy. Patients who have not had prior progression or grade 3 or greater toxicity with either daily temozolomide or etoposide or who have no prior exposure to either will be randomized to one of the groups. Bevacizumab will be administered intravenously at 10mg/kg every other week. Temozolomide will be administered ona continuous daily dosing schedule at 50 mg/m^2/day.
- Etoposide Arm: Bevacizumab + Etoposide: Patients who progressed or had grade 3 or greater toxicity related to prior daily temozolomide dosing, but have not had prior progression or grade 3 or greater toxicity related to prior daily etoposide therapy. Patients who have not had prior progression or grade 3 or greater toxicity with either daily temozolomide or etoposide or who have no prior exposure to either will be randomized to one of the groups. Bevacizumab will be administered intravenously at 10mg/kg every other week. Etoposide will be administered once daily at 50 mg/m^2/day for the first 21 days of each 28-day cycle.
Period: Overall Study
Arm/Group | Temozolomide Arm | Etoposide Arm
Started | 10 | 13
Completed | 10 | 12
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Temozolomide Arm: Pts treated w Bev + Temozolomide
- Etoposide Arm: Pts treated w Bev + Etoposide
- Total: Total of all reporting groups
Arm/Group | Temozolomide Arm | Etoposide Arm | Total
Number analyzed (Participants) | 10 | 13 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (9.1) | 51.7 (13.8) | 51.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is 6 Month Progression-free Survival.
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or to death due to any cause.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temozolomide Arm | Etoposide Arm
Number analyzed (Participants) | 10 | 13
percentage of participants | 0 [0 to 0] | 7.7 [4.8 to 29.2]

2. Secondary Outcome: Radiographic Response
Description: Percentage of participants with an objective response (complete response or partial response) based on modified Macdonald criteria.
Time Frame: 41 months
Measure: Number; unit: percentage of participants
Arm/Group | Temozolomide Arm | Etoposide Arm
Number analyzed (Participants) | 10 | 12
percentage of participants | 0 | 0

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to Macdonald criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: 41 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Temozolomide Arm | Etoposide Arm
Number analyzed (Participants) | 10 | 13
weeks | 4.1 [3.0 to 7.9] | 8.1 [4.1 to 12.0]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 41 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Temozolomide Arm | Etoposide Arm
Number analyzed (Participants) | 10 | 13
weeks | 12.6 [4.6 to 23.3] | 19 [11.0 to 25.7]

5. Secondary Outcome: Grade 3 or Greater, Treatment Related, Non-hematologic Toxicities.
Description: Incidence of ≥Grade 3 treatment related, non-hematologic toxicity
Time Frame: 41 months
Measure: Number; unit: participants
Arm/Group | Temozolomide Arm | Etoposide Arm
Number analyzed (Participants) | 10 | 13
participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 41 months
Description: Adverse events were gathered and assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, but were converted to CTCAE version 4.0 for entry into ClinicalTrials.gov
Arm/Group | Temozolomide Arm | Etoposide Arm
Serious Adverse Events (participants affected / at risk) | 4/10 | 2/13
Other Adverse Events (participants affected / at risk) | 4/10 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide Arm (N=10) | Etoposide Arm (N=13)
Death NOS (General disorders) | 2 | 1
Infections and infestations-Other, specify: Bilateral Abscess in groin (Infection with normal ANC) (Infections and infestations) | 1 | 0
Infections and infestations-Other, specify: Shingles (Infections and infestations) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide Arm (N=10) | Etoposide Arm (N=13)
Blurred vision (Eye disorders) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 2 | 5
Ataxia (Nervous system disorders) | 1 | 4
Cognitive disturbance (Nervous system disorders) | 2 | 2
Dysphasia (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 0 | 3
Memory impairment (Nervous system disorders) | 2 | 3
Peripheral motor neuropathy (Nervous system disorders) | 2 | 6
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2
Reproductive system and breast disorders-Other, specify: Sexual Dysfunction (Reproductive system and breast disorders) | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No